CLINICAL TRIAL: NCT05120193
Title: Treatment of Persistent Atrial Fibrillation With the Sphere-9 Mapping and Ablation Catheter and the Affera Mapping and Ablation System
Brief Title: Treatment of Persistent Atrial Fibrillation With Sphere-9 Catheter and Affera Mapping and Ablation System
Acronym: SPHERE Per-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP-00009
Record Dates: First submitted 2021-10-25; First posted 2021-11-15 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects will be blinded to treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Sphere-9 Catheter (Experimental): Sphere-9™ Mapping and Ablation Catheter; Affera Mapping System; Affera Ablation System
  Interventions: Device: Mapping and Ablation
- THERMOCOOL SMARTTOUCH SF (Active Comparator): THERMOCOOL SMARTTOUCH® SF Catheter; SMARTABLATE® System; CARTO® 3 System
  Interventions: Device: Mapping and Ablation

INTERVENTIONS:
Device: Mapping and Ablation — Minimally invasive catheter mapping and ablation procedure

SUMMARY:
This is a prospective, multicenter, randomized clinical evaluation of the Sphere-9 Mapping and Ablation Catheter with the Affera Mapping and Ablation System. Subjects will be randomly assigned 1:1 to receive treatment with either the Sphere-9 Mapping and Ablation Catheter and the Affera Mapping and Ablation System (investigational device) or the THERMOCOOL SMARTTOUCH® SF radiofrequency ablation catheter (control device).

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic PerAF documented by (1) a physician's note indicating symptoms consistent with AF sustained longer than 7 days but less than 12 months; AND either (2a) a 24-hour Holter documenting continuous AF within the past year OR (2b) two electrocardiograms (from any form of rhythm monitoring, including consumer devices) taken at least 7 days apart within the past year, each showing continuous AF.
2. Failure or intolerance of at least one Class I or III anti-arrhythmic drug (AAD).
3. Suitable candidate for catheter ablation.
4. Adults aged 18 - 80 years.
5. Willing and able to comply with all baseline and follow-up evaluations for the full length of the study.
6. Willing and able to provide informed consent.

Exclusion Criteria:

1. Continuous AF lasting for 12 months or longer.
2. AF secondary to electrolyte imbalance, thyroid disease, acute alcohol intoxication, or other reversible or non-cardiac cause.
3. Previous left atrial ablation or surgical procedure (including septal closure or left atrial appendage closure).
4. Valvular cardiac surgical/percutaneous procedure (e.g., ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve).
5. Any carotid stenting or endarterectomy.
6. Any cardiac procedure (surgical or percutaneous) or percutaneous coronary intervention within the 90 days prior to the initial procedure.
7. Coronary artery bypass graft (CABG) procedure within the 6 months prior to the initial procedure.
8. Awaiting cardiac transplantation or other cardiac surgery within the 12 months following the initial ablation procedure.
9. Presence of a permanent pacemaker, biventricular pacemaker, or any type of implantable cardiac defibrillator (with or without biventricular pacing function).
10. Documented thromboembolic event (stroke or transient ischemic attack) within 6 months (180 days) prior to the initial ablation procedure.
11. Documented left atrial thrombus on imaging.
12. History of blood clotting or bleeding abnormalities.
13. Any condition contraindicating chronic anticoagulation.
14. Myocardial infarction (MI) within the 3 months (90 days) prior to the initial procedure.
15. Body mass index >40 kg/m2.
16. Left atrial diameter >55 mm (anterioposterior).
17. Diagnosed atrial myxoma.
18. Left ventricular ejection fraction (EF) < 35%.
19. Uncontrolled heart failure or NYHA Class III or IV heart failure.
20. Rheumatic heart disease.
21. Hypertrophic cardiomyopathy.
22. Unstable angina.
23. Moderate to severe mitral valve stenosis.
24. Severe mitral regurgitation (regurgitant volume ≥ 60 mL/beat, regurgitant fraction ≥ 50%, and/or effective regurgitant orifice area ≥ 0.40cm2).
25. Primary pulmonary hypertension.
26. Significant restrictive or obstructive pulmonary disease or chronic respiratory condition.
27. Renal failure requiring dialysis.
28. History of severe Gastroesophageal Reflux Disease (GERD) requiring surgical and/or mechanical intervention.
29. Acute illness, active systemic infection, or sepsis.
30. Contraindication to both computed tomography and magnetic resonance angiography.
31. Significant congenital anomaly or medical problem that, in the opinion of the investigator, would preclude enrollment in this study or compliance with follow-up requirements or would impact the scientific soundness of the clinical study results.
32. Any woman known to be pregnant or breastfeeding, or any woman of childbearing potential who is not on a reliable form of birth regulation method or abstinence.
33. Current or anticipated participation in any other clinical study of a drug, device, or biologic during the duration of the study not pre-approved by the Sponsor.
34. Presence of intramural thrombus, tumor, or other abnormality that precludes vascular access, catheter introduction, or manipulation.
35. Known drug or alcohol dependency.
36. Life expectancy less than 12 months.
37. Vulnerable subject (such as a prisoner or handicapped or mentally disabled person).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (19):
  - Arrhythmia Institute at Grandview, Birmingham, Alabama
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Pacific Heart Institute, Santa Monica, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Naples Heart Institute, Naples, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Maimonides Medical Center, Brooklyn, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Northwell Health, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The OhioHealth Research Institute, Columbus, Ohio
  - Doylestown Hospital, Doylestown, Pennsylvania
  - University of Pittsburgh Medical Center Pinnacle Health, Wormleysburg, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Czechia (3):
  - Nemocnice Ceske Budejovice, České Budějovice
  - Institut Klinicke a Experimentani Mediciny, Prague
  - Nemocnice Na Homolce, Prague
- Shamir Medical Center, Zrifin, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mansour M, Sharma D, Kiehl EL, Nair DG, Neuzil P, Kautzner J, Osorio J, Natale A, Mountantonakis SE, Hummel JD, Amin AK, Doshi SK, Siddiqui UR, Cerkvenik J, van Bragt KA, Tarakji KG, Anter E, Reddy VY, Taigen TL; SPHERE Per-AF Investigators. Impact of linear ablation in persistent atrial fibrillation using a dual energy, wide-footprint catheter - Analysis from the SPHERE Per-AF Randomized Trial. Heart Rhythm. 2026 Feb 6:S1547-5271(26)00099-8. doi: 10.1016/j.hrthm.2026.01.037. Online ahead of print. PMID 41655663
- [Derived] Matsumoto K, van Bragt KA, Kueffer FJ, Mburu W, Tarakji KG. Indirect treatment comparison of two pulsed field ablation systems for the treatment of persistent atrial fibrillation. J Interv Card Electrophysiol. 2025 Sep 10. doi: 10.1007/s10840-025-02124-6. Online ahead of print. PMID 40928625
- [Derived] Kiehl EL, Mountantonakis SE, Mansour MC, Nair DG, Sharma D, Taigen TL, Neuzil P, Kautzner J, Osorio J, Natale A, Hummel JD, Amin AK, Siddiqui UR, Bulava A, Doshi SK, Patel CP, Greenberg YJ, Tung RH, Harlev D, Hultz P, Rosen S, van Bragt KA, Tarakji KG, Reddy VY, Anter E; SPHERE Per-AF Investigators. Operator learning curve with a novel dual-energy lattice-tip ablation system. Heart Rhythm. 2026 Jan;23(1):89-96. doi: 10.1016/j.hrthm.2025.02.006. Epub 2025 Feb 6. PMID 39922404
- [Derived] Anter E, Mansour M, Nair DG, Sharma D, Taigen TL, Neuzil P, Kiehl EL, Kautzner J, Osorio J, Mountantonakis S, Natale A, Hummel JD, Amin AK, Siddiqui UR, Harlev D, Hultz P, Liu S, Onal B, Tarakji KG, Reddy VY; SPHERE PER-AF Investigators. Dual-energy lattice-tip ablation system for persistent atrial fibrillation: a randomized trial. Nat Med. 2024 Aug;30(8):2303-2310. doi: 10.1038/s41591-024-03022-6. Epub 2024 May 17. PMID 38760584

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 37 Roll-In subjects, 8 subjects that exited the study prior to randomization, and 12 randomized subjects that exited the study prior to the index ablation procedure.
Groups:
- Sphere-9 Catheter: Sphere-9™ Catheter; Affera Mapping System; Affera Ablation System
  Mapping and Ablation: Minimally invasive catheter mapping and ablation procedure
Period: Overall Study
Arm/Group | Sphere-9 Catheter | THERMOCOOL SMARTTOUCH SF
Started | 212 | 208
Completed | 209 | 199
Not Completed | 3 | 9

BASELINE CHARACTERISTICS:
Population: Subjects who provided informed consent, were randomized and underwent insertion of the assigned study device (experimental or active comparator), defined as the device emerging from the sheath into the bloodstream.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sphere-9 Catheter | THERMOCOOL SMARTTOUCH SF | Total
Number analyzed (Participants) | 212 | 208 | 420
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 73 | 134
  >=65 years | 151 | 135 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (8.3) | 66.7 (8.8) | 67.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 61 | 134
  Male | 139 | 147 | 286
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 206 | 201 | 407
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 2 | 6
  White | 199 | 199 | 398
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 177 | 179 | 356
  Czechia | 32 | 26 | 58
  Israel | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With a Primary Adverse Event
Description: The primary safety endpoint is the incidence of the following device- or procedure-related serious adverse events (SAEs) following the index ablation procedure:
  Within 7 days:
  * Death
  * Myocardial infarction
  * Phrenic nerve paralysis
  * Transient ischemic attack (TIA)
  * Stroke/cerebrovascular accident (CVA)
  * Thromboembolism
  * Major vascular access complications / bleeding
  * Heart block
  * Gastroparesis
  * Severe pericarditis
  * Hospitalization due to cardiovascular or pulmonary AE
  Within 30 days:
  • Cardiac tamponade / perforation
  Within 90 days:
  • Atrio-esophageal fistula
  Within 180 days:
  • Pulmonary vein stenosis
Time Frame: 180 Days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sphere-9 Catheter | THERMOCOOL SMARTTOUCH SF
Number analyzed (Participants) | 212 | 208
Participants | 3 | 2
Statistical Analysis 1: Comparison: Sphere-9 Catheter vs THERMOCOOL SMARTTOUCH SF; The null hypothesis (H0) for the primary safety analysis is that the true rate of primary safety events for the investigational device (QI) is equal to or greater than the true rate for the control device (QC) plus a non-inferiority margin (NIM) of 0.08. The alternative hypothesis (HA) is that the rate of primary safety events for the investigational arm (QI) is less than the rate of primary safety events for the control arm (QC) plus the NIM of 0.08. H0: QI ≥ QC + 0.08 HA: QI < QC + 0.08; Test type: Non-Inferiority — The primary safety analysis is performed at a one-sided Type I error rate of α = 0.05. The Farrington-Manning method is used to calculate the upper 95% confidence bound for the difference (QI - QC) between the rate of the primary safety endpoint in the investigational arm (QI) and the rate of the primary safety endpoint in the control arm (QC). If the upper confidence bound is less than 0.08, the study is considered to have demonstrated safety of the investigational device; p < 0.0001, Farrington-Manning; Risk Difference (RD) = 0.005, 90% CI 2-sided [-0.028 to 0.037]

2. Primary Outcome: Percent of Subjects Free From Primary Effectiveness Failure
Description: The primary effectiveness endpoint is freedom from documented recurrence of AF, atrial tachycardia (AT), or atrial flutter (AFL) based on electrocardiographic data through 12-month follow-up and excluding a 90-day blanking period. The following are considered primary effectiveness endpoint failures:
  * Inability to isolate all targeted pulmonary veins during the index procedure.
  * Ablation using devices other than the assigned study device for any left atrial ablation during the index procedure.
  * Any repeat ablation, surgical ablation, or arrhythmia surgery for treatment of recurrent AF/AT/AFL after the index procedure.
  * Documented AF/AT/AFL recurrence after the 90-day blanking period.
  * Class I or III AAD dose increase from the historic maximum ineffective dose (prior to the index procedure) or initiation of a new Class I or III AAD for treatment of AF/AT/AFL after the 90-day blanking period.
  * DC cardioversion for AF/AT/AFL after the 90-day blanking period.
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sphere-9 Catheter | THERMOCOOL SMARTTOUCH SF
Number analyzed (Participants) | 210 | 202
Participants | 155 | 133
Statistical Analysis 1: Comparison: Sphere-9 Catheter vs THERMOCOOL SMARTTOUCH SF; The null hypothesis (H0) is that the true rate of primary effectiveness endpoint success (no failures through Day 360) for the investigational device (PI) is less than or equal to the true rate for the control device (PC) minus the NIM of 0.15. The alternative hypothesis (HA) is that the success rate for the investigational arm (PI) is greater than the success rate for the control device (PC) minus the NIM of 0.15. H0: PI ≤ PC - 0.15 HA: PI > PC - 0.15; Test type: Non-Inferiority — The primary effectiveness analysis (PSE) is performed at a one-sided Type I error rate of α = 0.025. The Farrington-Manning method is used to calculate the lower 97.5% confidence bound for the difference (PI - PC) between the rate of the PSE in the investigational arm (PI) and the rate of the PSE in the control arm (PC). If the lower confidence bound is greater than -0.15, the study is considered to have demonstrated effectiveness of the investigational device; p = 0.025, Farrington-Manning; Risk Difference (RD) = 0.08, 95% CI 2-sided [-0.009 to 0.168]

3. Secondary Outcome: Energy Application Time
Description: Total energy application time during the index ablation procedure
Time Frame: Day 0
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sphere-9 Catheter | THERMOCOOL SMARTTOUCH SF
Number analyzed (Participants) | 212 | 206
minutes | 7.1 (2.0) | 36.4 (17.7)
Statistical Analysis 1: Comparison: Sphere-9 Catheter vs THERMOCOOL SMARTTOUCH SF; The null hypothesis (H0) is that the mean total energy application time during the ablation procedure for the investigational device (ETI) is greater than or equal to the mean time for the control device (ETC). The alternative hypothesis (HA) is that the mean total energy application time for the investigational device is less. H0: ETI ≥ ETC versus HA: ETI < ETC; Test type: Superiority; p < 0.0001, t-test, 1 sided; Mean Difference (Final Values) = -29.2, 95% CI 2-sided [-31.7 to -26.8]

4. Secondary Outcome: Treatment Time
Description: Time from start to end of energy delivery
Time Frame: Day 0
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sphere-9 Catheter | THERMOCOOL SMARTTOUCH SF
Number analyzed (Participants) | 212 | 208
minutes | 46.7 (20.0) | 73.5 (34.4)
Statistical Analysis 1: Comparison: Sphere-9 Catheter vs THERMOCOOL SMARTTOUCH SF; The null hypothesis (H0) is that the mean treatment time for the investigational device (TTI) is greater than or equal to the mean treatment time for the control device (TTC). The alternative hypothesis (HA) is that the mean treatment time for the investigational device is less. H0: TTI ≥ TTC versus HA: TTI < TTC; Test type: Superiority; p < 0.0001, t-test, 1 sided; Mean Difference (Final Values) = -26.8, 95% CI 2-sided [-32.2 to -21.4]

5. Secondary Outcome: Procedure Time
Description: Time from start to end of venous access
Time Frame: Day 0
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sphere-9 Catheter | THERMOCOOL SMARTTOUCH SF
Number analyzed (Participants) | 212 | 208
minutes | 100.9 (30.8) | 126.1 (49.2)
Statistical Analysis 1: Comparison: Sphere-9 Catheter vs THERMOCOOL SMARTTOUCH SF; The null hypothesis (H0) is that the mean procedure time for the investigational device (PTI) is greater than or equal to the mean procedure time for the control device (PTC). The alternative hypothesis (HA) is that the mean procedure time for the investigational device is less. H0: PTI ≥ PTC versus HA: PTI < PTC; Test type: Superiority; p = 0.025, t-test, 1 sided; Mean Difference (Final Values) = -25.1, 95% CI 2-sided [-33.0 to -17.3]

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Sphere-9 Catheter | THERMOCOOL SMARTTOUCH SF
All-Cause Mortality (participants affected / at risk) | 2/212 | 3/208
Serious Adverse Events (participants affected / at risk) | 36/212 | 41/208
Other Adverse Events (participants affected / at risk) | 0/212 | 0/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sphere-9 Catheter (N=212) | THERMOCOOL SMARTTOUCH SF (N=208)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 3 (3) | 5 (6)
Atrial Flutter (Cardiac disorders) | 2 (2) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3) | 3 (3)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (4) | 2 (2)
Coronary artery disease (Cardiac disorders) | 4 (4) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 3 (3)
Thyroid disorder (Endocrine disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vascular insufficiency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal mucosa erythema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (3)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Systemic infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mouth Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery dissection (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatomegaly (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Immune system disorders) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical device implantation (Surgical and medical procedures) | 0 (0) | 1 (1)
Polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT05120193/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT05120193/SAP_001.pdf